CLINICAL TRIAL: NCT00001946
Title: A Comparison of Contrast Enhanced Magnetic Resonance Angiography (MRA) and Conventional Angiography in the Diagnosis of Atherosclerotic Disease: A Pilot Study
Brief Title: Comparison of Magnetic Resonance Angiography and Standard Angiography in Diagnosing Atherosclerosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 000028; 00-CC-0028
Record Dates: First submitted 2000-01-18; First posted 2000-01-19 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2002-09

CONDITIONS: Atherosclerosis
Keywords: Magnetic Resonance Angiography; Gadolinium; Suburban Hospital; Atherosclerosis
MeSH Terms: conditions — Atherosclerosis

INTERVENTIONS:
Procedure: Magnetic resonance angiography

SUMMARY:
This study will evaluate ways to improve magnetic resonance angiography (MRA) for diagnosing atherosclerosis (hardening and narrowing of the arteries).

MRA is a new method for looking at arteries and veins without standard angiography, which requires inserting a catheter into a blood vessel, injecting a contrast material, and obtaining X-ray images. Current MRA techniques, however, do not depict the lumen (cavity) of small vessels well enough to accurately determine the extent of their narrowing. This study will test image processing methods with the eventual goal of improving MRA accuracy to the point that it can replace X-ray catheter angiography for diagnosing atherosclerotic disease.

Patients with atherosclerosis who have had conventional angiography at Suburban Hospital in Bethesda, MD, may be considered for this study. They will be screened with a brief history and physical examination, and those enrolled will have a MRA scan within 72 hours of their conventional angiogram. For this procedure, a catheter is placed in a vein in the patient's arm and the patient lies on a table that slides into a magnetic resonance imaging (MRI) scanner-a large donut-shaped machine with a magnetic field. Surface coils-flexible, padded antennae used to improve the quality of the pictures-are wrapped around the patient's legs. At times during the scan, the patient is asked to hold his or her breath for several seconds, and a contrast material called gadolinium is injected through the catheter in the vein. This substance enhances the images of blood flow in the vessels. The procedure generally takes about an hour and a half, although the actual imaging takes only a small part of that time.

DETAILED DESCRIPTION:
Contrast Enhanced Magnetic Resonance Angiography (MRA) is a developing technology for the non-invasive evaluation of arterial and venous structures which does not require x-ray based catheter angiography. While dramatic progress in MRA has recently been made, there are still substantial limitations in the accuracy of MRA in grading stenoses and detecting small accessory vessels. The purpose of this study is to recruit patients with documented atherosclerotic disease as confirmed on catheter angiography performed at Suburban Hospital for evaluation with state-of-the-art MRA on MRI units, also at Suburban Hospital. We intend to test new surface coils, new pulse sequence designs, and advanced image processing algorithms in order to improve MRA accuracy to the point that a large-scale study of MRA vs. conventional angiography is possible. The goal of this pilot study is to improve MRA to the point that it can reliably replace diagnostic x-ray catheter angiography in the evaluation of patients with atherosclerotic disease.

ELIGIBILITY:
Patient must be willing to participate in the study.

Patient must have documented atherosclerotic disease of an extracranial vessel by angiography performed within 72 hours of the MRA.

Patient must be referred by a physician who is caring for the patient and to whom the results will be provided.

Patient must be clinically stable and be judged by their physician able to tolerate lying in the MR gantry for up to 1.5 hours.

Patient must have serum Creatinine value less than 3.0mg/dl.

Must not have any contraindication for MRI including: pacemaker or other implanted electronic device; cochlear implants; metal in the eye; embedded shrapnel fragments; cerebral aneurysm clips; or medical Infusion pumps.

Must not have an allergy to Gadolinium based contrast media.

Must not have unsatisfactory performance status as judged by the referring physician such that the patient could not tolerate an MRI scan for 1.5 hours. Examples of medical conditions that would not be accepted would include unstable angina, dyspnea at rest, severe pain at rest, and severe back pain.

Must not have intercurrent illness that requires treatment that would be jeopardized by the MRA scan.

Subjects must not require sedation for MRI studies other than administered normally for a conventional angiogram.

Must not be pregnant.

Must not be nursing mothers.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Start 1999-12; Study Completion 2002-09

CONTACTS AND LOCATIONS:
Locations (1):
- Warren G. Magnuson Clinical Center (CC), Bethesda, Maryland, United States

REFERENCES:
- [Background] Prince MR, Yucel EK, Kaufman JA, Harrison DC, Geller SC. Dynamic gadolinium-enhanced three-dimensional abdominal MR arteriography. J Magn Reson Imaging. 1993 Nov-Dec;3(6):877-81. doi: 10.1002/jmri.1880030614. PMID 8280977
- [Background] Prince MR. Peripheral vascular MR angiography: the time has come. Radiology. 1998 Mar;206(3):592-3. doi: 10.1148/radiology.206.3.9494471. No abstract available.
- [Background] Prince MR. Contrast-enhanced MR angiography: theory and optimization. Magn Reson Imaging Clin N Am. 1998 May;6(2):257-67. PMID 9560485